CLINICAL TRIAL: NCT03969849
Title: A Two-Part, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Effects of a Single Dose of REGN5713-5714-5715 in Healthy Adult Subjects
Brief Title: Study to Assess the Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Effects of a Single Dose of REGN5713-5714-5715 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R5713-5714-5715-HV-1857; 2018-004681-34 (EudraCT Number)
Record Dates: First submitted 2019-05-28; First posted 2019-05-31 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Healthy Volunteers; Birch Pollen Allergy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Part A: Cohort 1 (Experimental): Part A: Cohort 1 randomized 3:1 will receive REGN5713-5714-5715 or matching placebo
  Interventions: Drug: REGN5713-5714-5715; Drug: Matching placebo
- Part A: Cohort 2 (Experimental): Part A: Cohort 2 randomized 3:1 will receive REGN5713-5714-5715 or matching placebo
  Interventions: Drug: REGN5713-5714-5715; Drug: Matching placebo
- Part A: Cohort 3 (Experimental): Part A: Cohort 3 randomized 3:1 will receive REGN5713-5714-5715 or matching placebo
  Interventions: Drug: REGN5713-5714-5715; Drug: Matching placebo
- Part A: Cohort 4 (Experimental): Part A: Cohort 4 randomized 3:1 will receive REGN5713-5714-5715 or matching placebo
  Interventions: Drug: REGN5713-5714-5715; Drug: Matching placebo
- Part B (Experimental): Part B: Randomized 1:1 will receive REGN5713-5714-5715 or matching placebo in Healthy Participants with birch pollen allergy
  Interventions: Drug: REGN5713-5714-5715; Drug: Matching placebo

INTERVENTIONS:
Drug: REGN5713-5714-5715 — Part A: Cohort 1 - 3: Single sequential ascending subcutaneous (SC) dose Part A: Cohort 4: Single intravenous (IV) dose Part B: Single SC dose
Drug: Matching placebo — Part A: Cohort 1 - 3: Single sequential ascending subcutaneous (SC) dose Part A: Cohort 4: Single intravenous (IV) dose Part B: Single SC dose

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of REGN5713-5714-5715 in healthy adult participants.

The secondary objectives of the study are:

In Part A and Part B:

* To characterize the concentration time profile of single doses of REGN5713-5714-5715 in healthy adults
* To assess the immunogenicity of single dose of REGN5713-5714-5715.

In Part B:

* To assess the inhibition of allergic symptoms as measured by total nasal symptom score (TNSS) provoked by a birch allergen nasal allergen challenge (NAC) in birch-sensitized allergic subjects after a single subcutaneous (SC) dose of REGN5713-5714-5715
* To assess the skin test reactivity provoked by a skin prick test (SPT) with serial birch allergen titration after a single SC dose of REGN5713-5714-5715.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant is judged by the investigator to be in good health based on medical history, physical examination, vital sign measurements, and ECG performed prior to study drug dosing
* Participant is in good health based on laboratory safety testing obtained at the screening prior to study drug dosing
* Part B: Has a medical history of birch tree pollen-triggered allergic rhinitis (AR) symptoms with or without conjunctivitis (for at least 2 seasons) based on participant's recall
* Part B: Has positive skin prick test (SPT) with birch tree pollen extract (mean wheal diameter ≥5 mm greater than a negative control) in screening period

Key Exclusion Criteria:

* History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric, or neurological disease, as assessed by the investigator that may confound the results of the study or pose an additional risk to the participant by study participation
* Has any physical examination findings and/or history of any illness that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the participant by study participation
* Participation in any clinical research study evaluating another investigational drug or therapy within 90 days or at least 5 half-lives (whichever is longer) for an investigational biologic drug, or at least 28 days for other investigational products, or within 6 months for immunotherapy prior to the screening visit of the current trial
* Pregnant or breastfeeding women
* Part B: Receipt of study drug REGN5713-5714-5715 in Part A
* Part B: Significant rhinitis or sinusitis outside of the birch pollen season or due to daily contact with other allergens causing symptoms, that is expected to coincide with the study NAC assessments as assessed by the investigator
* Part B: A clinical history of asthma requiring chronic medication such as regular, inhaled corticosteroids for >6 months per year
* Part B: History of birch allergy immunotherapy (SCIT, sublingual immunotherapy, or oral immunotherapy) in the 5 years prior to screening

NOTE: Other protocol defined inclusion/exclusion criteria apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-03-27 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) | Up to 16 Weeks
The number of participants with abnormal adverse events (AEs) | Up to 16 Weeks
The number of participants with abnormal vital signs | Up to 16 Weeks
  Vital signs include blood pressure, heart rate, body temperature, and respiratory rate
The number of participants with abnormal 12-lead electrocardiograms (ECGs) | Up to 16 Weeks
The number or participants with abnormal physical examinations | Up to 16 Weeks
  The limited physical examination will include assessment of heart, lungs, abdomen, peripheral pulses, and skin
The number of abnormal laboratory examination | Up to 16 Weeks
  Hematology, chemistry, urinalysis and pregnancy testing samples will be analyzed
Part B only - The number of participants with abnormal lung function using spirometry - forced vital capacity (FVC) litres (L) | Up to 16 Weeks
  Spirometry will be measured only in participants with a history of asthma prior to the NAC procedure. FVC is the total amount of air exhaled during the forced expiratory volume (FEV) test
Part B only - The number of participants with abnormal lung function using spirometry - forced expiratory volume in 1 second (FEV1) | Up to 16 Weeks
  Spirometry will be measured only in participants with a history of asthma prior to the NAC procedure. FEV in 1 second (FEV1) must be ≥80% predicted to perform the NAC. FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation
Part B only - The number of participants with abnormal lung function using spirometry - FEV1/FVC (%) | Up to 16 Weeks
  Spirometry will be measured only in participants with a history of asthma prior to the NAC procedure. FEV1 must be ≥80% predicted to perform the NAC.
Part B only - The number of participants with abnormal lung function using spirometry - peak expiratory flow (PEF) Litre/second (L/s) | Up to 16 Weeks
  Spirometry will be measured only in participants with a history of asthma prior to the NAC procedure. PEF is the maximum speed of expiration.
Part B only - The number of participants with abnormal lung function using spirometry - forced expiratory flow 25 to 75 (L/s) | Up to 16 Weeks
  Spirometry will be measured only in participants with a history of asthma prior to the NAC procedure. Forced expiratory flow during the mid (25 - 75%) portion of the FVC.
Part B only - The number of participants with poorly controlled asthma using asthma control test (ACT) | Up to 16 Weeks
  Performed prior to every NAC procedure in all participants. A multiple-choice questionnaire for patients with asthma, each choice is assigned a score 1-5. There are 5 questions to answer. The total score is calculated, ranging between 5 and 25. Lower scores indicate worse asthma control. Participants must have ACT ≥20 before undergoing the NAC.

SECONDARY OUTCOMES:
Total concentration of REGN5713 in serum over time | Up to 16 Weeks
Total concentration of REGN5714 in serum over time | Up to 16 Weeks
Total concentration of REGN5715 in serum over time | Up to 16 Weeks
Immunogenicity as measured by anti-drug antibodies (ADA) to REGN5713 | Up to 16 Weeks
Immunogenicity as measured by ADA to REGN5714 | Up to 16 Weeks
Immunogenicity as measured by ADA to REGN5715 | Up to 16 Weeks
Change in area under the curve (AUC) for TNSS (0 to 1 hour post-peak TNSS) in response to a nasal allergen challenge (NAC) from the pretreatment baseline TNSS AUC (0 to 1 hour post-peak TNSS) for REGN5713-5714-5715 as compared to placebo | At day 8, 29 and 57
Percent change in AUC for TNSS (0 to 1 hour post-peak TNSS) in response to a NAC from the pretreatment baseline TNSS AUC (0 to 1 hour post-peak TNSS) for REGN5713-5714-5715 as compared to placebo | At day 8, 29 and 57
Change in mean wheal diameters of the skin prick test with serial birch allergen titration from the pretreatment baseline for REGN5713-5714-5715 as compared to placebo | At day 8, 29 and 57
Percent change in mean wheal diameters of the skin prick test with serial birch allergen titration from the pretreatment baseline for REGN5713-5714-5715 as compared to placebo | At day 8, 29 and 57

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (3):
- Belgium (3):
  - Regeneron Study Site, Antwerp
  - Regeneron Study Site, Ghent
  - Regeneron Study Site, Leuven

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

REFERENCES:
- [Derived] Gevaert P, De Craemer J, De Ruyck N, Rottey S, de Hoon J, Hellings PW, Volckaert B, Lesneuck K, Orengo JM, Atanasio A, Kamal MA, Abdallah H, Kamat V, Dingman R, DeVeaux M, Ramesh D, Perlee L, Wang CQ, Weinreich DM, Herman G, Yancopoulos GD, O'Brien MP. Novel antibody cocktail targeting Bet v 1 rapidly and sustainably treats birch allergy symptoms in a phase 1 study. J Allergy Clin Immunol. 2022 Jan;149(1):189-199. doi: 10.1016/j.jaci.2021.05.039. Epub 2021 Jun 11. PMID 34126156